CLINICAL TRIAL: NCT01189149
Title: Intravenous Fluids vs. Naso/Orogastric-tube Feeding in Hospitalized Infants With Acute Viral Bronchiolitis: a Randomized, Controlled, Prospective Clinical Trial
Brief Title: Intravenous Fluids Versus Naso/Orogastric-tube Feeding in Hospitalized Infants With Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115/08
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2009-12

CONDITIONS: Viral Bronchiolitis
MeSH Terms: conditions — Bronchiolitis, Viral | interventions — Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV fluids (Experimental): Infants will get IV fluids whem indicated until able to tolerate full oral feedings
  Interventions: Procedure: IV fluids
- Oro/naso gastric tube feeding (Experimental): Infants will get oro/naso gastric tube feeding whem indicated until able to tolerate full oral feedings
  Interventions: Procedure: Naso/oro gastric tube feedings

INTERVENTIONS:
Procedure: IV fluids — Infants will be allocated to IV fluids
  Arms: IV fluids
Procedure: Naso/oro gastric tube feedings — Infants will be allocated to naso/oro gastric tube feedings
  Arms: Oro/naso gastric tube feeding

SUMMARY:
Oro- or nasogastric tube feeding is safe and may be more physiologic than intravenous (IV) fluids in hospitalized infants with acute viral bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Infants with bronchiolitis < 6 months who need to be hospitalized and are not able to eat per os.

Exclusion Criteria:

* Infants with severe bronchiolitis not allowed to get any gastric feeds or those that their parents will not sign an informed consent.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | 3 winters
  Will compare clinical outcomes between the groups: Length of stay, need for oxygen, time to full feeds etc.

SECONDARY OUTCOMES:
Possible side effects of each method (IV vs. Oro/nasogastric feedings) | 3 winters
  Local or systemic signs of infection, "para"infusion, discomfort while inserting the IV, electrolyte abnormalitis (as part of routine care) vs. aspiration, discomfort with naso/oro gastric tube.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kugelman, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Pediatric Department, Haifa, Israel

REFERENCES:
- [Derived] Kugelman A, Raibin K, Dabbah H, Chistyakov I, Srugo I, Even L, Bzezinsky N, Riskin A. Intravenous fluids versus gastric-tube feeding in hospitalized infants with viral bronchiolitis: a randomized, prospective pilot study. J Pediatr. 2013 Mar;162(3):640-642.e1. doi: 10.1016/j.jpeds.2012.10.057. Epub 2012 Dec 20. PMID 23260101